CLINICAL TRIAL: NCT05539131
Title: Demonstration Study of the Effect of the Transcranial Direct Current Stimulation (tDCS) for the Patients With Depression in Clinical Fields
Brief Title: Demonstration Study of the Effect of the Transcranial Direct Current Stimulation (tDCS) on Depressed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Woo Jung Kim, Clinical Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0225-002
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active transcranial direct current stimulation (tDCS) (Active Comparator): daily active transcranial direct current stimulation (tDCS) use for 6 weeks
  Interventions: Device: transcranial direct current stimulation (tDCS)
- sham transcranial direct current stimulation (tDCS) (Sham Comparator): daily active transcranial direct current stimulation (tDCS) use for 3 weeks + daily sham transcranial direct current stimulation (tDCS) use for 3 weeks
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation (tDCS) suppresses excitability and regulates excitability of neurons by injecting a small amount of current through electrodes attached to the scalp.

SUMMARY:
Purpose of research: It aims to demonstrate the effectiveness of transcranial direct current stimulation (tDCS) in the clinical domain for patients with depression and to optimize home-based e-medication technology.

DETAILED DESCRIPTION:
As a home-based clinical empirical study of transcranial direct current stimulation for depressed patients, male and female subjects aged 19 to 65 who meet the criteria for mild and moderate Major depressive disorder (MDD) were enrolled, and real-world data (RWD) was obtained through self-application of transcranial direct current stimulation (tDCS) at home for 6 weeks. This is a study that secures and derives real-world evidence (RWE) that can be applied to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged 19 to 65 with mild and moderate Major depressive disorder (MDD)

Exclusion Criteria:

* Those diagnosed with Post-traumatic stress disorder (PTSD), Obsessive compulsive disorder (OCD), bipolar or psychotic major depressive disorder, high suicide risk, Electroencephalography (EEG) and DC stimulation electrode attachment problems (such as scalp deformity, inflammatory response or other dermatological problems), Transcranial direct current stimulation (tDCS) medical device taboos (such as head metal plate insertion), clinical trials that have been inadequate for clinical trials

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Woo Jung Kim, Principal Investigator — Severance Hospital
Locations (5):
- South Korea (5):
  - Hallym Univsity Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - National Health Insurance Service Ilsanhospital, Goyang-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Catholic Kwandong University International St. Mary'S Hospital, Incheon, Gyeonggi-do
  - Yongin Severance Hospital, Yonsei University College of Medicine, Yongin, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Yes
Personal information collected for research purposes shall be kept anonymously in a safe place within the institute to be managed so that personal information is not exposed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the completion of the study, the data will be available for 3 years.
Access Criteria: For data security, encrypted communication methods will be used and restricted access to only authorized licensed personnel on the e-CRF domain.
URL: https://console.redea.io/

REFERENCES:
- [Background] Oh J, Jang KI, Jeon S, Chae JH. Effect of Self-administered Transcranial Direct Stimulation in Patients with Major Depressive Disorder: A Randomized, Single-blinded Clinical Trial. Clin Psychopharmacol Neurosci. 2022 Feb 28;20(1):87-96. doi: 10.9758/cpn.2022.20.1.87. PMID 35078951
- [Background] Fregni F, Nitsche MA, Loo CK, Brunoni AR, Marangolo P, Leite J, Carvalho S, Bolognini N, Caumo W, Paik NJ, Simis M, Ueda K, Ekhitari H, Luu P, Tucker DM, Tyler WJ, Brunelin J, Datta A, Juan CH, Venkatasubramanian G, Boggio PS, Bikson M. Regulatory Considerations for the Clinical and Research Use of Transcranial Direct Current Stimulation (tDCS): review and recommendations from an expert panel. Clin Res Regul Aff. 2015 Mar 1;32(1):22-35. doi: 10.3109/10601333.2015.980944. PMID 25983531
- [Background] Wang J, Luo H, Schulke R, Geng X, Sahakian BJ, Wang S. Is transcranial direct current stimulation, alone or in combination with antidepressant medications or psychotherapies, effective in treating major depressive disorder? A systematic review and meta-analysis. BMC Med. 2021 Dec 17;19(1):319. doi: 10.1186/s12916-021-02181-4. PMID 34915885
- [Derived] Park HY, Park J, Roh D, Jhung K, Chang JG, Park S, Ryu JS, Do G, Lee K, Park JY, Kim WJ. Real-World Effects of Home-Based Transcranial Direct Current Stimulation in Depression: A Randomized Controlled Trial of 3-Week Versus 6-Week Protocols. Brain Behav. 2025 Dec;15(12):e71119. doi: 10.1002/brb3.71119. PMID 41376187

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Before assignment to study arms, 12 participants were excluded during the screening phase due to failure to meet eligibility criteria (e.g., comorbid psychiatric conditions or contraindications to tDCS).
Groups:
- Active (Real): Participants received 6 weeks of active transcranial direct current stimulation (tDCS) at 2 mA, 5 days per week.
- Sham: Participants received 3 weeks of active tDCS followed by 3 weeks of sham stimulation (placebo control).
Period: Overall Study
Arm/Group | Active (Real) | Sham
Started | 108 | 89
Completed | 89 | 57
Not Completed | 19 | 32

BASELINE CHARACTERISTICS:
Population: Active (Real) tDCS Group: Participants received 6 weeks of active transcranial direct current stimulation (tDCS) treatment at 2 mA, 5 days per week.
  Sham tDCS Group: Participants received 3 weeks of active tDCS treatment followed by 3 weeks of sham stimulation (placebo control).
Groups:
- Active (Real): Participants received 6 weeks of active transcranial direct current stimulation (tDCS) treatment at 2 mA, 5 days per week.
- Sham: Participants received 3 weeks of active tDCS treatment followed by 3 weeks of sham stimulation (placebo control).
- Total: Total of all reporting groups
Arm/Group | Active (Real) | Sham | Total
Number analyzed (Participants) | 108 | 89 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 108 | 89 | 197
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 51 | 124
  Male | 35 | 38 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 108 | 89 | 197
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 108 | 89 | 197
Beck Depression Inventory-II(BDI-II) [Mean (Standard Deviation); unit: units on a scale] — It is a self-report depression scale of 21 questions, which the score range from 0 to 63, and it is required to select a sentence that is appropriate for you among 4 descriptions for each question, and the total score is 0 to 63 points for each question. 0~13: Minimal 14~19: Mild depression 20~28: Moderate depression 29~63: Severe depression
  units on a scale | 30.27 (13.22) | 29.62 (11.12) | 30.00 (12.35)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depressive Symptoms on Beck Depression Inventory-II (BDI-II) at Week 13
Description: It is a self-report depression scale of 21 questions, which the score range from 0 to 63, and it is required to select a sentence that is appropriate for you among 4 descriptions for each question, and the total score is 0 to 63 points for each question.
  0~13: Minimal 14~19: Mild depression 20~28: Moderate depression 29~63: Severe depression
Time Frame: From Visit1(baseline) to 91 days
Population: Eligible individuals were adults aged 19-65 years with a primary diagnosis of mild to moderate MDD, as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (Association, 2013) and confirmed using the Mini International Neuropsychiatric Interview (Sheehan et al., 1998).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active (Real): 6WA, 6-week active stimulation.
- Sham: 3WA, 3-week active followed by 3-week sham stimulation.
Arm/Group | Active (Real) | Sham
Number analyzed (Participants) | 108 | 89
units on a scale
  Visit1(Baseline) | 30.27 (13.22) | 29.62 (11.12)
  Visit2(18~24 days from the baseline): number analyzed (Participants) | 98 | 65
  Visit2(18~24 days from the baseline) | 24.96 (13.01) | 23.98 (13.32)
  Visit3(39~45 days from the baseline): number analyzed (Participants) | 89 | 57
  Visit3(39~45 days from the baseline) | 24.35 (13.85) | 22.09 (13.66)
  Visit4(77~91 days from the baseline): number analyzed (Participants) | 77 | 55
  Visit4(77~91 days from the baseline) | 22.81 (14.9) | 20.49 (14.46)
Statistical Analysis 1: Comparison: Active (Real) vs Sham; Test type: Superiority — The LMM analysis results refer to the F-statistics and associated p-values derived from linear mixed-effects models (LMMs), including fixed effects for time, group, and their interaction; p = 0.862, Mixed Models Analysis — This is p-valu regarding time and group

2. Primary Outcome: Change From Baseline in Depressive Symptoms on Montgomery-Asberg Depression Rating Scale (MADRS) at Week 13
Description: It evaluates 10 items such as apparent sadness, voluntarily reporting sadness, internal tension, sleep loss, loss of appetite, laziness, loss of feeling, pessimistic thinking, and suicide accident, and the total score is 0 to 60 points per question.
  It evaluates 10 items such as apparent sadness, voluntarily reporting sadness, internal tension, sleep loss, loss of appetite, laziness, loss of feeling, pessimistic thinking, and suicide accident, and the total score is 0 to 60 points per question.
  It evaluates 10 items such as apparent sadness, voluntarily reporting sadness, internal tension, sleep loss, loss of appetite, laziness, loss of feeling, pessimistic thinking, and suicide accident, and the total score is 0 to 60 points per question.
  The total score ranges from 0 to 60 points. 0-6 indicate an absence of symptoms 7-19 Mild depression 20-34 Moderate depression 35-60 Severe depression
Time Frame: From Visit1(baseline) to 91 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active (Real) | Sham
Number analyzed (Participants) | 108 | 89
units on a scale
  Visit1(Baseline) | 25.63 (8.15) | 24.29 (7.71)
  Visit2(18~24 days from the baseline): number analyzed (Participants) | 98 | 65
  Visit2(18~24 days from the baseline) | 19.76 (8.40) | 19.43 (8.79)
  Visit3(39~45 days from the baseline): number analyzed (Participants) | 89 | 57
  Visit3(39~45 days from the baseline) | 19.15 (9.26) | 18.42 (10.91)
  Visit4(77~91 days from the baseline): number analyzed (Participants) | 77 | 55
  Visit4(77~91 days from the baseline) | 19.30 (10.35) | 17.13 (12.95)
Statistical Analysis 1: Comparison: Active (Real) vs Sham; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.662, Mixed Models Analysis — This is p-valu regarding time and group

3. Secondary Outcome: Change From Baseline in Depressive Symptoms on Epidemiologic Studies Depression Scale Revised (CESD-R) at Week 13
Description: Epidemiologic Studies Depression Scale Revised test was revised to reflect the major depressive illustration diagnostic criteria for the evaluation of depression. Items reflecting anaesthesia, mental exercise delay/anxiety, and suicide accidents have been added, and are measured as 0 to 4 points per question on a self-report 20 question scale. The score ranges from 0~80 points. . A score equal to or above 16 indicates a person at risk for clinical depression.
Time Frame: From Visit1(baseline) to 91 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active (Real) | Sham
Number analyzed (Participants) | 108 | 89
units on a scale
  Visit1(Baseline) | 36.83 (17.74) | 36.40 (16.37)
  Visit2(18~24 days from the baseline): number analyzed (Participants) | 98 | 65
  Visit2(18~24 days from the baseline) | 34.39 (17.86) | 31.53 (19.15)
  Visit3(39~45 days from the baseline): number analyzed (Participants) | 89 | 57
  Visit3(39~45 days from the baseline) | 30.73 (18.42) | 26.25 (19.39)
  Visit4(77~91 days from the baseline): number analyzed (Participants) | 77 | 55
  Visit4(77~91 days from the baseline) | 27.19 (18.95) | 23.84 (19.06)
Statistical Analysis 1: Comparison: Active (Real) vs Sham; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.318, ANOVA — This is p-valu regarding time and group

4. Secondary Outcome: Change From Baseline in Depressive Symptoms on Hamilton Anxiety Scale (HAM-A) at Week 13
Description: The scale developed by Hamilton consists of 14 questions, and is evaluated by the clinician on a 5-point Likert scale of a semi-structured interview tool. The score ranges from 0~56 points. Each item is scored on a scale of 0 (not present) to 4 (severe), with total score range of 0-56, where <17 indi- cates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: From Visit1(baseline) to 91 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active (Real) | Sham
Number analyzed (Participants) | 108 | 89
units on a scale
  Visit1(Baseline) | 16.22 (9.01) | 17.44 (7.67)
  Visit2(18~24 days from the baseline): number analyzed (Participants) | 98 | 65
  Visit2(18~24 days from the baseline) | 13.18 (8.07) | 14.62 (9.09)
  Visit3(39~45 days from the baseline): number analyzed (Participants) | 89 | 57
  Visit3(39~45 days from the baseline) | 13.70 (9.49) | 13.11 (8.70)
  Visit4(77~91 days from the baseline): number analyzed (Participants) | 77 | 55
  Visit4(77~91 days from the baseline) | 12.92 (8.99) | 13.15 (10.48)
Statistical Analysis 1: Comparison: Active (Real) vs Sham; Test type: Superiority; p = 0.273, ANOVA

5. Secondary Outcome: Change From Baseline in Depressive Symptoms on Clinical Global Impression-Severity of Illness Scale (CGI-SI) at Week 13
Description: It was developed for evaluation of symptom severity, treatment response, and treatment effectiveness in patients with psychiatric disorders (Guy W, 1976) and scored 0-7 points based on the overall impression of the subject's symptoms and treatment response compared to typical patients with the disease.
  It was developed for evaluation of symptom severity, treatment response, and treatment effectiveness in patients with psychiatric disorders (Guy W, 1976) and scored 0-7 points based on the overall impression of the subject's symptoms and treatment response compared to typical patients with the disease. The score ranges from 0~7 points. 1: normal, not at all ill 2: borderline mentally ill 3: mildly ill 4: moderately ill 5: markedly ill 6: severely ill 7: extremely ill
Time Frame: From Visit1(baseline) to 91 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active (Real) | Sham
Number analyzed (Participants) | 108 | 89
units on a scale
  Visit1(Baseline) | 3.19 (1.01) | 3.35 (0.89)
  Visit2(18~24 days from the baseline): number analyzed (Participants) | 98 | 65
  Visit2(18~24 days from the baseline) | 2.87 (0.94) | 3.04 (1.02)
  Visit3(39~45 days from the baseline): number analyzed (Participants) | 89 | 57
  Visit3(39~45 days from the baseline) | 2.74 (1.04) | 2.95 (1.11)
  Visit4(77~91 days from the baseline): number analyzed (Participants) | 77 | 55
  Visit4(77~91 days from the baseline) | 2.75 (1.11) | 2.75 (1.13)
Statistical Analysis 1: Comparison: Active (Real) vs Sham; Test type: Superiority; p = 0.639, ANOVA

6. Secondary Outcome: Change From Baseline in Depressive Symptoms on Digit Symbol Substitution Test (DSST) at Week 13
Description: t is possible to measure high-dimensional cognitive functions such as perceptual organization ability and visual movement coordination, and examine attentional concentration, visual short-term memory, and mental movement speed. A post-marketing survey (PMS) on a new mechanism of anti-depressant (vortioxetine) is used to measure cognitive function before and after the use of the antidepressant in depressed patients. The score is the number of correct number-symbol matches achieved in 90 s. The score ranges from 0~93 points.
Time Frame: From Visit1(baseline) to 91 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active (Real) | Sham
Number analyzed (Participants) | 108 | 89
units on a scale
  Visit1(Baseline) | 42.39 (11.45) | 42.09 (11.12)
  Visit2(18~24 days from the baseline): number analyzed (Participants) | 98 | 65
  Visit2(18~24 days from the baseline) | 46.58 (11.39) | 46.78 (9.98)
  Visit3(39~45 days from the baseline): number analyzed (Participants) | 89 | 57
  Visit3(39~45 days from the baseline) | 48.83 (11.67) | 48.95 (10.59)
  Visit4(77~91 days from the baseline): number analyzed (Participants) | 77 | 55
  Visit4(77~91 days from the baseline) | 49.51 (12.10) | 48.09 (10.54)
Statistical Analysis 1: Comparison: Active (Real) vs Sham; Test type: Superiority; p = 0.452, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were systematically collected over a mean of 13 weeks during the 6-week intervention period and the follow-up visit immediately following the end of the study.
Description: Adverse event information was collected using systematic assessments, including standardized questionnaires, regular investigator assessments, and participant self-reports during study visits. The definition of adverse events aligns with clinicaltrials.gov guidelines, focusing on events temporally associated with study participation, regardless of causality.
Groups:
- Active: 6WA, 6-week active stimulation.
- Sham(1): 3-week active followed
- Sham(2): 3-week sham stimulation.
Arm/Group | Active | Sham(1) | Sham(2)
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/89 | 0/89
Serious Adverse Events (participants affected / at risk) | 2/108 | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 3/108 | 5/89 | 1/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=108) | Sham(1) (N=89) | Sham(2) (N=89)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=108) | Sham(1) (N=89) | Sham(2) (N=89)
Skin irriation (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT05539131/Prot_SAP_000.pdf